CLINICAL TRIAL: NCT06786624
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NBI-1065845 as Adjunctive Treatment in Subjects With Major Depressive Disorder (MDD)
Brief Title: Study to Assess the Efficacy and Safety of NBI-1065845 as an Adjunctive Treatment in Participants With Major Depressive Disorder (MDD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065845-MDD3024; 2024-519418-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Major Depressive Disorder; NBI-1065845; TAK-653; MADRS
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-1065845 (Experimental): NBI-1065845 administered orally once a day.
  Interventions: Drug: NBI-1065845
- Placebo (Placebo Comparator): Placebo identical in appearance to NBI-1065845 will be administered orally once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1065845 — NBI-1065845 tablets
  Other Names: TAK-653
  Arms: NBI-1065845
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of NBI-1065845 compared with placebo as an adjunctive treatment in participants with MDD on improving symptoms of depression.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of recurrent MDD (moderate or severe) or persistent depressive disorder.
* Participant has had an inadequate response to oral antidepressant treatments in the current episode of depression.
* Participant must have been taking oral antidepressants for at least 8 weeks and is willing to continue the same oral antidepressants at the same dose and frequency of administration throughout participation in the study.
* Total Hamilton Depression Rating Scale-17 Item (HAM-D17) score ≥22 at screening and at study baseline (Day 1).
* Willing and able to comply with all study procedures and restrictions in the opinion of the investigator.

Key Exclusion Criteria:

* A current or prior psychiatric disorder diagnosis in the last 1 year that was the primary focus of treatment other than MDD.
* Are considered by the investigator to be at imminent risk of suicide or injury to self or others.
* Participants depressive symptoms have previously demonstrated nonresponse to electroconvulsive therapy (ECT) in the current major depressive episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Montgomery-Åsberg Depression Rating Scale (MADRS) Score at Day 56 | Baseline, Day 56

SECONDARY OUTCOMES:
Change from Baseline in Sheehan Disability Scale (SDS) Total Score at Day 56 | Baseline, Day 56
Change from Baseline in Clinical Global Impression-Severity Scale (CGI-S) Score at Day 56 | Baseline, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (18):
- United States (18):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Garden Grove, California
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Upland, California
  - Neurocrine Clinical Site, Hollywood, Florida
  - Neurocrine Clinical Site, Maitland, Florida
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Watertown, Massachusetts
  - Neurocrine Clinical Site, Mount Kisco, New York
  - Neurocrine Clinical Site, Avon Lake, Ohio
  - Neurocrine Clinical Site, Westlake, Ohio
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Richmond, Texas
  - Neurocrine Clinical Site, The Woodlands, Texas
  - Neurocrine Clinical Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No